CLINICAL TRIAL: NCT02760082
Title: Identifying Motivational Factors for Registering Nutrition and Lifestyle Factors Among Patients With Multiple Sclerosis
Brief Title: Motivation of Patients Diagnosed With Multiple Sclerosis to Become Citizen Researchers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Multiple Sclerosis Society (Unknown)
Responsible Party: Principal Investigator, Astrid Knudsen, Industrial PhD Student, University of Copenhagen
Other Study IDs: 12016SCL
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Qualitative study; Motivation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Semi-structured interviews: 20 participants (anticipated)
  Interventions: Other: Qualitative evaluation
- Questionnaire survey: 400 respondents (anticipated)
  Interventions: Other: Qualitative evaluation
- Focus group interviews: 3-5 focus group interviews (anticipated)
  Interventions: Other: Qualitative evaluation

INTERVENTIONS:
Other: Qualitative evaluation

SUMMARY:
The study will based on qualitative methods investigate motivational factors among patients diagnosed with multiple sclerosis for registering nutrition, environmental factors, stress provoking factors and physical activity (NESPA). The aim is to gain knowledge on motivational factors for using a digital tool for collecting data on NESPA and incorporate this knowledge into a form which can be used in requirement specifications for such a digital tool.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Read, write and understand Danish

Exclusion Criteria:

* Aphasia
* Severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Multiple Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Analysis of qualitative interviews and measurement of eHealth literacy (eHealth literacy questionnaire) | Up to 6 months
Evaluation of motivational factors based on questionnaire survey | Up to 10 months
Analysis of focus group interviews on motivational factors for registering nutrition and lifestyle factors among patients with multiple sclerosis | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No